CLINICAL TRIAL: NCT04158401
Title: Cervical Stiffness Measurement in Cervical Insufficiency
Status: Completed | Type: Observational
Sponsor: Tufts Medical Center (Other)
Collaborators: Pregnolia AG (Industry)
Responsible Party: Sponsor
Other Study IDs: 13549
Record Dates: First submitted 2019-10-23; First posted 2019-11-08 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Pregnancy Related; Cervical Insufficiency; Preterm Birth
MeSH Terms: conditions — Uterine Cervical Incompetence; Premature Birth

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Control group: Pregnant patients between 12w0d and 22w0d who present for prenatal care.
  Interventions: Device: Pregnolia
- Cerclage group A: Patients who present for a history-indicated cerclage placement.
  Interventions: Device: Pregnolia
- Cerclage group B: Patients who present for an ultrasound-indicated cerclage placement.
  Interventions: Device: Pregnolia
- Cerclage group C: Patients who present for an exam-indicated cerclage placement.
  Interventions: Device: Pregnolia

INTERVENTIONS:
Device: Pregnolia — The Pregnolia measurement device (CE Mark for commercialization in the EU) will be used to measure the cervical stiffness (Pcl) on all subjects.

SUMMARY:
The goal of this cross sectional study is to evaluate the differences in cervical stiffness between patients who present for cerclage placement versus normal pregnancies.

The central hypothesis is that women for whom a cerclage is indicated will have cervical stiffness measurements lower than normal controls. Cervical stiffness will be objectively measured by the closing pressure Pcl using the Pregnolia measurement device. This is performed during a speculum exam by placing the measurement probe on the ectocervix.

In current clinical care, there is no objective measurement of cervical stiffness. An accurate measurement of cervical stiffness that correlates with clinical outcome will advance the field. Successful completion of the current study will spark future studies that correlate cervical stiffness pcl in a prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women over 18 years of age.
2. Singleton gestation.
3. Gestational ages between 12w0d and 22w6d.
4. Candidates for cerclage
5. Normal controls, which will be matched to cerclage subjects by gestational age and parity

Exclusion Criteria:

1. Multiple gestation pregnancy.
2. Pregnancy complications: Premature rupture of membranes, Placental abruption, Placenta previa/accreta.
3. Chorioamnionitis
4. Preterm contractions
5. History of cervical surgery (LEEP, trachelectomy, conization).
6. Mullarian anomaly
7. Known carrier or HIV or Hepatitis B/C
8. Active genital infection
9. Communication problems (cognitively impaired adults unable to give consent)
10. Cerclage placement already performed this pregnancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Patients need to be pregnant.
Study Population: We are studying pregnant patients between 12w0d and 22w6d.
Sampling Method: Non-Probability Sample
Enrollment: 136 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2022-06-15 (Actual); Study Completion 2022-06-15 (Actual)

PRIMARY OUTCOMES:
Cervical stiffness (Pcl) | 5 minutes
  The primary outcome will be cervical stiffness, Pcl in patients presenting for cerclage versus normal controls.

SECONDARY OUTCOMES:
Delivery data | up to 10 months
  Patient delivery data including gestational age, mode of delivery and complications will be recorded
Newborn outcomes | up to 10 months
  Newborn outcomes including weight, APGARs and complications will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Michael House, MD, Principal Investigator — Tufts Medical Center
Locations (1):
- Tufts Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lorenz JM. The outcome of extreme prematurity. Semin Perinatol. 2001 Oct;25(5):348-59. doi: 10.1053/sper.2001.27164. PMID 11707021
- [Background] Goldenberg RL, Culhane JF, Iams JD, Romero R. Epidemiology and causes of preterm birth. Lancet. 2008 Jan 5;371(9606):75-84. doi: 10.1016/S0140-6736(08)60074-4. PMID 18177778
- [Background] Gilbert WM, Nesbitt TS, Danielsen B. The cost of prematurity: quantification by gestational age and birth weight. Obstet Gynecol. 2003 Sep;102(3):488-92. doi: 10.1016/s0029-7844(03)00617-3. PMID 12962929
- [Background] Iams JD, Johnson FF, Sonek J, Sachs L, Gebauer C, Samuels P. Cervical competence as a continuum: a study of ultrasonographic cervical length and obstetric performance. Am J Obstet Gynecol. 1995 Apr;172(4 Pt 1):1097-103; discussion 1104-6. doi: 10.1016/0002-9378(95)91469-2. PMID 7726247
- [Background] Beck S, Wojdyla D, Say L, Betran AP, Merialdi M, Requejo JH, Rubens C, Menon R, Van Look PF. The worldwide incidence of preterm birth: a systematic review of maternal mortality and morbidity. Bull World Health Organ. 2010 Jan;88(1):31-8. doi: 10.2471/BLT.08.062554. Epub 2009 Sep 25. PMID 20428351
- [Background] Mazza E, Parra-Saavedra M, Bajka M, Gratacos E, Nicolaides K, Deprest J. In vivo assessment of the biomechanical properties of the uterine cervix in pregnancy. Prenat Diagn. 2014 Jan;34(1):33-41. doi: 10.1002/pd.4260. PMID 24155152
- [Background] Hollenstein M, Bugnard G, Joos R, Kropf S, Villiger P, Mazza E. Towards laparoscopic tissue aspiration. Med Image Anal. 2013 Dec;17(8):1037-45. doi: 10.1016/j.media.2013.06.001. Epub 2013 Jun 19. PMID 23876854
- [Background] Badir S, Bajka M, Mazza E. A novel procedure for the mechanical characterization of the uterine cervix during pregnancy. J Mech Behav Biomed Mater. 2013 Nov;27:143-53. doi: 10.1016/j.jmbbm.2012.11.020. Epub 2012 Dec 11. PMID 23274486
- [Background] Badir S, Mazza E, Zimmermann R, Bajka M. Cervical softening occurs early in pregnancy: characterization of cervical stiffness in 100 healthy women using the aspiration technique. Prenat Diagn. 2013 Aug;33(8):737-41. doi: 10.1002/pd.4116. Epub 2013 Apr 29. PMID 23553612
- [Background] Bauer M, Mazza E, Jabareen M, Sultan L, Bajka M, Lang U, Zimmermann R, Holzapfel GA. Assessment of the in vivo biomechanical properties of the human uterine cervix in pregnancy using the aspiration test: a feasibility study. Eur J Obstet Gynecol Reprod Biol. 2009 May;144 Suppl 1:S77-81. doi: 10.1016/j.ejogrb.2009.02.025. Epub 2009 Mar 13. PMID 19285777
- [Background] Bauer M, Mazza E, Nava A, Zeck W, Eder M, Bajka M, Cacho F, Lang U, Holzapfel GA. In vivo characterization of the mechanics of human uterine cervices. Ann N Y Acad Sci. 2007 Apr;1101:186-202. doi: 10.1196/annals.1389.004. Epub 2007 Mar 15. PMID 17363446
- [Background] Mazza E, Nava A, Bauer M, Winter R, Bajka M, Holzapfel GA. Mechanical properties of the human uterine cervix: an in vivo study. Med Image Anal. 2006 Apr;10(2):125-36. doi: 10.1016/j.media.2005.06.001. Epub 2005 Sep 6. PMID 16143559
- [Background] Mazza E, Nava A, Hahnloser D, Jochum W, Bajka M. The mechanical response of human liver and its relation to histology: an in vivo study. Med Image Anal. 2007 Dec;11(6):663-72. doi: 10.1016/j.media.2007.06.010. Epub 2007 Jul 5. PMID 17719834
- [Background] ACOG Practice Bulletin No.142: Cerclage for the management of cervical insufficiency. Obstet Gynecol. 2014 Feb;123(2 Pt 1):372-379. doi: 10.1097/01.AOG.0000443276.68274.cc. PMID 24451674